CLINICAL TRIAL: NCT00033176
Title: Immune Restoration by Lipoic Acid in AIDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT000246-01A2 (NIH)
Record Dates: First submitted 2002-04-08; First posted 2002-04-09 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: complementary therapies; Immune restoration; HIV infection; AIDS; HAART non-responsiveness; glutathione restoration; lipoic acid; dithiol
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Thioctic Acid

INTERVENTIONS:
Drug: Alpha Lipoic Acid

SUMMARY:
The purpose of this study is to determine the immunomodulatory and antiviral effects of the glutathione-restoring dithiol, alpha lipoic acid (ALA) in HIV-infected persons unresponsive to highly active antiretroviral treatment (HAART).

DETAILED DESCRIPTION:
AIDS is characterized by infection with HIV which leads to collapse of the immune system. Although highly active antiretroviral therapy (HAART) has contributed significantly to lowering morbidity and mortality from AIDS, antiretroviral drugs do not fully restore the immune system and patients often fail multi-drug treatment. Hence, there is a need for alternative/complementary medicine (CAM) that can restore an immune system ravaged by HIV/AIDS. To address this need, investigators have formed a multidisciplinary collaboration to evaluate and demonstrate utility of natural immune-based modulators in ethnically diverse patients with HIV/AIDS. The long-term goal of this proposal is to develop a CAM therapy to facilitate immune reconstitution and HIV eradication following cessation of antiretroviral treatment or concurrent with continued antiretroviral treatment. It is based on the premise of a widespread deficiency of glutathione (GSH), vital to lymphocyte function, in patients with HIV/AIDS. The proposed project will study the immunomodulatory and antiretroviral effects of a dietary antioxidant, alpha-lipoic acid (ALA), which is known to efficiently boost systemic GSH.

In this study, HIV-infected adults unresponsive to HAART (i.e. those with persistent CD4+ count > 50 cells/mm3, viral load> 10,000 copies/cc) will be randomized into a treatment or a control arm. The treatment group will be given 300 mg ALA thrice daily for 6 months and the control group will receive inert placebo. Studies performed at baseline and at 2,4, and 6 months will include estimation of CD4+ count, HIV RNA, T-cell reactivity in vitro and whole blood GSH level. Significance of changes from baseline parameters will be analyzed by t-tests. The proposed research will show whether GSH augmentation by ALA increases CD4+ cell number and T cell function and reduces viral load in subjects unresponsive to antiretroviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive status
* HAART non-responsiveness as defined by 1) previous experience with at least 2 different protease inhibitors plus nucleoside analogs; 2) viral load of >10,000 copies/cc and CD4+ cell count >50 x 1000 cells/liter at time of enrollment

Exclusion Criteria:

* Diabetic patients
* Pregnant women
* Asthmatic patients
* Severely thiamine-deficient persons (e.g. alcoholics and those with polyneuritis)
* History of supplementing on excessive amounts of N-acetylcysteine, glutathione or other antioxidant supplements, during the 2 months prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33
Dates: Start 2002-02; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Raxit J. Jariwalla, PhD, Principal Investigator — California Institute for Medical Research; Abha Kumar, MD — Santa Clara Valley Medical Center; Jay Lalezari, MD — Quest Clinical Research
Locations (2):
- United States (2):
  - Quest Clinical Research, San Francisco, California
  - Eye Clinic, Santa Clara Valley Medical Center, San Jose, California